CLINICAL TRIAL: NCT01685086
Title: Surveillance and Follow-up for Latent Tuberculosis Infection and Observation of the Effect of Prophylactic Latent Tuberculosis Treatment in Patients With Severe Chronic Kidney Disease or Receiving Long-term Dialysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201110013RC
Record Dates: First submitted 2012-09-11; First posted 2012-09-13 (Estimated); Last update posted 2012-09-13 (Estimated); Status verified 2011-11

CONDITIONS: To Determine the Prevalence of Latent Tuberculosis in Each Group; To Monitor the Occurrence of Active Tuberculosis
Keywords: latent tuberculosis infection, tuberculosis, chronic kidney disease, peritoneal dialysis, hemodialysis
MeSH Terms: conditions — Latent Tuberculosis; Tuberculosis; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Patients with severe chronic kidney disease
- Patient with peritoneal dialysis
- Patients with hemodialysis

SUMMARY:
To follow-up the latent tuberculosis infection and evaluate the risk of developing active tuberculosis in patients with severe chronic kidney disease or receiving long-term dialysis

DETAILED DESCRIPTION:
Tuberculosis (TB) remains an important infectious disease worldwide. Taiwan is still an edemic area. In 2008, there is an incidence of 62 persons having TB per 100,000 population. To control TB, we should prevent further TB transmission via early diagnosis and treatment of latent TB. In screening the risk population for TB, patients with renal failure acquiring long-term dialysis, in addition to close contacts, have higher incidence and mortality than general population. Moreover, the risk for active TB in dialysis patients is ten to 25 times larger. In Taiwan, the dialysis group is important because it has higher prevalence (2228 per in per million people by 2009 annual report of United States Renal Data System) than other countries in the world. In particular, the dialysis patients usually has an extrapulmonary presentation for their TB, so diagnosis is always delay. Hence, we should detect latent TB in those dialysis patients for monitor them from active tuberculosis.

Currently, interferon-gamma release assays (IGRAs) are used for finding out those with latent TB and have been proven useful for those being immunocompromised, and having BCG vaccination. For dialysis patients, IGRAs have been tested and been considered better than skin tuberculin test. However, previous studied rarely observed the patients receiving peritoneal dialysis and severe chronic kidney disease. Besides, those cross-sectional studies used the indirect evidence for diagnosis and lacked longitudinal follow-up. We thus conducted this study for observing the prevalence of latent TB in those receiving hemodialysis or peritoneal dialysis by using IGRAs. We also kept follow-up for the primary outcome of active TB occurrence.

ELIGIBILITY:
Inclusion Criteria:

* older than 20 years old
* Estimated CCr < 30 ml/min as group of severe chronic kidney disease
* Long-term (>3months) dialysis as dialysis group

Exclusion Criteria:

* refusal of recruitment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with severe chronic kidney disease or long term dialysis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-03

PRIMARY OUTCOMES:
occurrence of active tuberculosis | 2 years

SECONDARY OUTCOMES:
Latent tuberculosis infection | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Chung Shu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan